CLINICAL TRIAL: NCT04301869
Title: Oral Versus Intravenous Antibiotics for the Treatment of Pleural Space Infection: a Randomized Controlled Pilot Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Vaibhav Mokashi (Unknown)
Responsible Party: Principal Investigator, Phillipe El-Helou, Principal Investigator, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSI Trial
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Pleural Infection
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous therapy (Active Comparator): Intravenous antibiotics administered for pleural space infection
  Interventions: Drug: Antibiotics
- Oral therapy (Active Comparator): Oral antibiotics administered for pleural space infection
  Interventions: Drug: Antibiotics

INTERVENTIONS:
Drug: Antibiotics — Oral versus intravenous therapy

SUMMARY:
We aim to conduct a pilot trial assessing oral versus intravenous therapy for pleural space infections.

DETAILED DESCRIPTION:
Pleural space infections are a frequent clinical problem resulting in significant morbidity and mortality as well as healthcare cost. Despite the increasing burden of disease, there are no clinical trials evaluating antibiotic therapy in pleural space infections. Hence, British and American guidelines are only able to provide weak and vague recommendations regarding duration, type or route (intravenous or oral) of antibiotic therapy. Our goal is to determine whether oral (PO) therapy is non-inferior to intravenous (IV) therapy thereby decreasing risks of IV catheter related infections, vein thrombosis and health care costs. Similar studies have been successfully conducted in the setting of bone/joint infections and endocarditis and showed non-inferiority of oral antibiotics. However, in order to help ensure that the randomized trial is of good quality, it is important to assess the feasibility of such a trial by first conducting a pilot study. The goal of this pilot trial is to assess the feasibility of the proposed study design.

ELIGIBILITY:
Inclusion Criteria:

* Must meet our study definition of pleural space infection
* Age > or = 18 years old
* Life expectancy > 1 year
* Received intravenous or oral antibiotics for = or < 7 d from surgical intervention or received a total of = or < 7 d of antibiotics if no intervention performed

Exclusion Criteria:

* S. aureus bacteremia or endocarditis in the last 1 month
* Another concomitant infection requiring prolonged IV antibiotics
* Esophageal rupture or malignant pleural effusion
* Septic shock or systemic features requiring IV antibiotics
* Mycobacterial, fungal or parasitic pleural space infection
* No oral antibiotic options available
* Unlikely to comply with therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Enrollment feasibility | 3 months
  Proportion of eligible participants screened that are randomized within 5 days of initial intravenous antibiotic exposure
Completion feasibility | 3 months
  Proportion of participants with follow-up at 4 weeks either through a clinic visit or phone call

SECONDARY OUTCOMES:
Treatment failure | 3 months
  Treatment failure at the 3-month clinical visit or phone conversation, defined as any of: (i) return to the emergency department for new fever, shortness of breath or progressive hypoxia OR (ii) radiological progression of empyema or development of a new abscess OR (iii) mortality related to pleural space infection. Treatment failure must be agreed upon by the majority of the adjudication committee.
Mortality | 3 months
  All-cause mortality at 3 months
Antibiotic duration | 3 months
  Duration of antibiotics with start date as the date of randomization
Hospitalization duration | 3 months
  Duration of hospitalization
Stopping antibiotics | 3 months
  Early termination of antibiotics due to patient intolerance, patient preference or any other reason.
IV line complications | 3 months
  Infection, thrombosis or new line placement for IV catheter-related issues.
C. difficile | 3 months
  Clostridium difficile associated diarrhea as per the accepted PIDAC definition

IPD SHARING:
Plan to Share IPD: Undecided